CLINICAL TRIAL: NCT02004002
Title: Dietary Protein Intake, Insulin Sensitivity and β-cell Function
Brief Title: Protein Intake & Insulin Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSP-201303080
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight maintenance with normal protein intake (Active Comparator): Control group will consume 1.4 g protein/kg body wt/d; consistent with the average protein intake in the US population.
  Interventions: Behavioral: Weight maintenance with normal protein intake
- Weight maintenance with protein restriction (Experimental): Protein restriction group will receive the Institute of Medicine RDA of 0.8 g protein/kg body wt/d.
  Interventions: Behavioral: Weight maintenance with protein restriction

INTERVENTIONS:
Behavioral: Weight maintenance with normal protein intake — Control group will consume 1.4 g/kg/d of protein; consistent with the average protein intake in the US population.
  Arms: Weight maintenance with normal protein intake
Behavioral: Weight maintenance with protein restriction — Protein restriction group will receive the Institute of Medicine RDA of 0.8 g protein/kg body wt/d.
  Arms: Weight maintenance with protein restriction

SUMMARY:
The purpose of this proposal is to determine whether dietary protein restriction has beneficial effects on skeletal muscle insulin sensitivity and β-cell function in obese men and women.

DETAILED DESCRIPTION:
Insulin resistance, impaired pancreatic β-cell function, and diabetes are important complications associated with obesity. Although excess energy intake and body fat accumulation are considered the major culprits responsible for obesity-associated metabolic abnormalities, it is possible that insulin resistance and impaired β-cell function are also due to increased dietary protein intake.

Protein intake is ~15 to 25% greater in obese than lean adults and exceeds the current Institute of Medicine Recommended Daily Allowance (RDA) of 0.8 g protein/kg body weight by ~75%. An increase in habitual protein intake of only 10 to 40%, assessed using dietary recall methods, been shown to increase the risk of developing diabetes by up to 2.2 fold. Additionally, the ability to stimulate glucose disposal during insulin infusion is reported to be impaired in individuals consuming double the recommended protein intake as part of an isoenergetic diet. However, it is not known whether decreasing protein intake can improve insulin sensitivity and β-cell function in weight-stable, obese individuals.

Accordingly, obese men and women will be randomized to 8 weeks of treatment with a weight maintaining diet containing either i) 0.8 g protein/kg body weight (as recommended by the Institute of Medicine; protein restriction group)or ii) 1.4 g protein/kg body weight (control group). All subjects will receive a standardized "base-diet" with or without protein supplementation to avoid potential food selection bias that could confound the results when using high- and low-protein diets.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 30 and 50 kg/m2
* Subjects who are sedentary (<1.5 h of exercise/week)
* Subjects with a high habitual protein intake (>1.2 g/kg body mass/day)

Exclusion Criteria:

* Subjects with evidence of significant organ system dysfunction (e.g. diabetes, severe cardiovascular disease, hyperlipidemia, cirrhosis, hypogonadism, uncontrolled hypo- or hyperthyroidism; uncontrolled hypertension)
* Subjects with metal implants
* Individuals with cancer or cancer that has been in remission for <5 years,
* Individuals with dementia,
* Individuals who use tobacco products,
* Subjects who are taking medications known to affect glucose metabolism (e.g., steroids),
* Subjects taking medications to control certain medical conditions (e.g., hypertension) will be included if the drug regimen has been stable for at least 6 months before entering the study and is not expected to change during the study.
* Women who are pregnant due to changes in body composition and decreases in insulin sensitivity caused by pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | up to 8 wk dietary intervention
  We will evaluate insulin sensitivity using the hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotope labeled tracer infusions.
total β-cell sensitivity index (Φtotal) | Before and after the 8 wk dietary intervention
  The total β-cell sensitivity index assesses the insulin secretion response to changes in plasma glucose concentration following ingestion of a glucose drink.

SECONDARY OUTCOMES:
Disposition index | Before and after the 8 wk dietary intervention
  The disposition index provides an assessment of insulin secretion in relationship to insulin sensitivity to determine whether insulin secretion was "appropriate" for the degree of insulin sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Smith, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States